CLINICAL TRIAL: NCT06054009
Title: Treating 'Felt Sense of Anomaly'-Type Dissociative Experiences by Targeting Hypothesised Psychological Maintenance Mechanisms: A Single Case Experimental Design Series
Brief Title: Dissociation CBT Studies
Acronym: DisCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RG_23-015; 325448 (Other: IRAS); 23/NW/0163 (Other: NHS Research Ethics Committee)
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-11

CONDITIONS: Dissociation; Depersonalization; Dissociative Disorder
Keywords: 'felt sense of anomaly'
MeSH Terms: conditions — Dissociative Disorders; Depersonalization

STUDY DESIGN:
Intervention Model Description: Three N=4 randomised multiple baseline design (MBD) single case experimental design studies, with A1B1A2 structure.
Masking Description: This study does not involve blinding. However, to incorporate a degree of impartiality, assessments will be carried out by a research assistant, not the therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): In Study 1: x4 CBT sessions addressing cognitive appraisals of dissociation. In Study 2: x4 CBT sessions addressing rumination/worry. In Study 3: x4 CBT sessions addressing affect intolerance.
  Interventions: Behavioral: Brief CBT

INTERVENTIONS:
Behavioral: Brief CBT — In Study 1: x4 CBT sessions addressing cognitive appraisals of dissociation. In Study 2: x4 CBT sessions addressing rumination/worry. In Study 3: x4 CBT sessions addressing affect intolerance.
  Other Names: CBT

SUMMARY:
Dissociation involves distressing feelings of unreality and disconnection. Evidence suggests it is particularly common amongst people with existing mental health difficulties, where it has been linked with greater clinical severity, poorer treatment response, and increased self-harm and suicidality. However, there are currently no psychological treatments for dissociation that have been developed from a scientific understanding of its underpinning psychological factors.

In this project, three studies, each with four participants, will test a different psychological factor. Participants will be: adults (16+ years); on a waiting list for NHS psychological therapy; high scorers on a dissociation questionnaire. Participants will complete assessments before and after treatment, and at a one-month follow-up. The studies follow a 'multiple baseline design', meaning that all four participants for that study will complete their baseline assessment in the same week, and then be randomly allocated to wait either one, two, three, or four weeks before starting the intervention. The intervention will consist of four therapy sessions taking place within a five-week 'window'. Taking part in the research is voluntary. Before deciding whether to participate, we will explain the study and answer any questions.

Daily, participants will record a score for their dissociation and the psychological factor being targeted. At baseline, post-therapy, and follow-up, the researchers will also measure their levels of other factors related to dissociation (i.e. those not targeted by the therapy). Additionally, feedback will be requested from participants about the therapy at the end of their involvement, in order to improve it in future.

Ultimately, if successful, these interventions could form a pilot therapy for further testing and development. This could mean fewer people struggle with the challenges of dissociation.

DETAILED DESCRIPTION:
1. What is dissociation?

   "I was in a totally different world; it was going on all around me. I thought that I might have died and was in hell, and I was thinking maybe that's what it was." -- "Maria"

   Dissociation involves confusing and upsetting feelings of unreality, unfamiliarity, or disconnection in relation to your mind, body, or surroundings. For example, some people describe being detached from their own emotions, including affection for loved ones, or feeling profoundly 'strange', as though they are living life from behind a thick pane of glass. These experiences can cause significant distress, and have been linked with risk of self-harm or suicide, and with increased severity and incomplete treatment-response of comorbid mental health diagnoses. Many dissociative experiences considered transdiagnostic. For example, dissociation is present at a very high rate in psychotic disorders (potentially up to 50%). Crucially, in this context, it may even be instrumental in the development and maintenance of key psychotic symptoms, such as paranoid delusions and auditory hallucinations.

   However, dissociation has traditionally been considered within the context of post-traumatic responses. As a result, a fuller understanding of dissociation as an independent construct - rather than simply as another post-traumatic symptom - has yet to be achieved.

   This 'neglect', and extensive debate within the field, has also resulted in a lack of clarity about the precise accepted definition of 'dissociation' as a construct. Therefore, in previous work, our research group delineated a subgroup of common dissociative experiences unified by a core phenomenological experience of a 'felt sense of anomaly' (FSA). Thus, the term 'dissociation' is operationalised within this project by focusing on this specific type of dissociative experiences (FSA-dissociation), since this has been demonstrated to be common and transdiagnostic.
2. What are the psychological maintenance mechanisms of dissociation?

   Understanding the psychological mechanisms of a pathological presentation is vital to developing an effective intervention for it. Seminal work developing (now gold standard) cognitive behavioural therapy (CBT) interventions for anxiety disorders and PTSD have demonstrated the clinical efficacy of identifying, verifying, and then precisely targeting the underlying causal mechanisms of the problem to be treated. However, much remains unknown about the psychological mechanisms underpinning dissociation. To date, only two experimental studies inferring causality in dissociation have been carried out: one of which was by our group.

   In our recent work, we began the process of identifying plausible mechanisms of FSA-dissociation, resulting in a provisional cognitive model of the problem. This model suggests that dissociative experiences are maintained by a two feedback loops. The first is caused by catastrophic appraisals (negative interpretations or beliefs about the dissociative experience), which lead to rumination and counterproductive 'safety behaviours' (actions intended to mitigate potential harm), both of which serve to keep attention focused on the dissociation and reinforce interpretations of this experience as threatening. This first loop therefore proposes three possible maintenance mechanisms: catastrophic appraisals of dissociation, perseverative thinking (rumination), and counterproductive safety behaviours.

   The second hypothesised feedback loop explains why the appraisals of dissociation are catastrophic in nature - as opposed to benign or benevolent. Across two large studies of online survey and NHS patient (psychosis) respondents, previous data has indicated relationships between dissociation and both high affect intolerance and low self-efficacy. In essence, people who feared shifts or peaks in their mood, and simultaneously felt powerless to manage or cope with challenges, were more likely to have FSA-dissociative experiences - as was indicated by previous qualitative evidence. This second feedback loop therefore suggests two further plausible mechanisms of dissociation: affect intolerance and self-efficacy.

   In this project, the researchers have chosen to focus on the three mechanisms with the largest effect sizes from this research: negative cognitive appraisals of the dissociative experience (causal effect 0.73 in a non-clinical group; 0.72 in a psychosis group), perseverative thinking (rumination) (0.31; 0.52), and affect intolerance (0.26; 0.41).
3. The current study

The aim of this project is therefore to test the three largest psychological contributors to FSA-dissociation as identified in this previous research: cognitive appraisals, rumination, and affect intolerance. Whilst there is evidence that these are all associated with dissociative experiences in the context of psychosis, to date there has been no experimental manipulation of these factors to demonstrate their role in maintaining dissociative difficulties. Evidence of their causal effect on dissociation is required before a translational psychological intervention can be developed.

Using an interventionist-causal approach (experimentally manipulating the factor of interest via attempting to ameliorate it with therapeutic techniques) allows researchers to combine an experimental test of causal relationships with the first stages of treatment development. This project constitutes an intermediate stage along the trajectory of treatment development, in that the primary aim of these three studies will be to demonstrate proof-of-concept for the interventions, in order that a larger study with adequate statistical power to test for causal relationships and treatment efficacy may be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16 years to 80 years;
* Outpatient of UK mental health services (at the time of referral to the study);
* Experiencing significant levels of 'felt sense of anomaly'-type dissociation (defined as a score within the 'moderately severe' or 'severe' range on the ČEFSA-14 (i.e., 39 or above); Černis et al., in prep.);
* Want help to improve their dissociative experiences;
* Willing and able to give consent for participation in the study;
* Available to undertake the baseline assessment in the indicated week;
* Available to undertake the therapy sessions within the indicated therapy 'window'.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Diagnosis of an Axis II ("personality") disorder;
* Primary diagnosis of alcohol/substance dependency, organic syndrome, or learning disability;
* Presence of risk issues that would be a clinical priority above managing dissociative symptoms (e.g., moderate to severe self-harm; active suicidal behaviour; etc.);
* Current engagement in any other individual psychological therapy (or psychological therapy due to begin within the participation window for this study).
* A participant may also not enter the study if there is another factor (i.e., with higher clinical priority), which, in the judgement of the investigator, would preclude the participant from providing informed consent or from safely engaging with the study procedures.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Study 1: Cognitive Appraisals of Dissociation | Through study completion, average of 3 months
  Visual Analogue Scale (0-100 rating) for cognitive appraisals of dissociation (higher scores = worse outcome)
Study 2: Perseverative Thinking | Through study completion, average of 3 months
  Visual Analogue Scale (0-100 rating) for cognitive appraisals of perseverative thinking (higher scores = worse outcome)
Study 3: Affect intolerance | Through study completion, average of 3 months
  Visual Analogue Scale (0-100 rating) for affect intolerance (higher scores = worse outcome)

SECONDARY OUTCOMES:
Levels of dissociative experience (felt sense of anomaly subtype dissociation) | Through study completion, average of 3 months
  Visual Analogue Scale (0-100 rating) for FSA-dissociation (higher scores = worse outcome)

OTHER OUTCOMES:
Acceptability of therapy and study to participants | Through study completion, average of 3 months
  Qualitative feedback (written or verbal)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Cernis, DPhil, Principal Investigator — University of Birmingham
Locations (1):
- Birmingham Womens and Childrens NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample sizes of each of the three studies, individual data will not be shared.

REFERENCES:
- See also: Open Science Framework project page, including pre-registered protocol — https://doi.org/10.17605/OSF.IO/RWC9N

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT06054009/Prot_SAP_001.pdf